CLINICAL TRIAL: NCT01462630
Title: Phase II Study Evaluating the Role of Pazopanib in Angiosarcoma
Brief Title: Pazopanib Hydrochloride in Treating Patients With Advanced Angiosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAR-043; NCI-2011-01314 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-042 (Other: Fox Chase Cancer Center); OER-SAR-043 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-07

CONDITIONS: Adult Angiosarcoma; Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Hemangiosarcoma; Sarcoma | interventions — pazopanib; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive pazopanib hydrochloride PO QD. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pazopanib hydrochloride; Other: laboratory biomarker analysis; Procedure: positron emission tomography; Procedure: computed tomography; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Drug: pazopanib hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Other: laboratory biomarker analysis — Correlative studies
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Correlative studies
  Other Names: tomography, computed
Radiation: fludeoxyglucose F 18 — Correlative studies
  Other Names: 18FDG; FDG

SUMMARY:
This phase II trial studies how well pazopanib hydrochloride works in treating patients with advanced angiosarcoma. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression free survival (PFS) at 3 months and response rate defined as complete response (CR) and partial response (PR) in angiosarcoma patients treated with pazopanib.

SECONDARY OBJECTIVES:

I. To assess overall survival of patients treated with pazopanib. II. To gather more safety data for pazopanib in this patient population. III. To explore the ability of [F-18] fludeoxyglucose (FDG) (positron emission tomography [PET])/computed tomography (CT) imaging to assess response.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up

  * Note: informed consent may be obtained prior to start of the specified screening window
  * Note: procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study such as bone scan) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
* Histologically or cytologically proven diagnosis of advanced stage angiosarcoma that is not amenable to treatment with curative intent; specify site of origin as cutaneous vs. non-cutaneous
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Must have measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 or cutaneous disease amenable to serial measurements should be present; a measurable lesion is defined as a lesion that can be accurately measured in at least one dimension with the longest diameter >= 10 mm with computed tomography (CT) scan; lesions that have been treated with therapeutic intent will be considered measurable if they have increased in size by more than 20%
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Hemoglobin >= 9 g/dL (5.6 mmol/L)
* Platelets >= 100 X 10^9/L
* International normalized ratio (INR) =< 1.2 X upper limit of normal (ULN)
* Activated partial thromboplastin time (aPTT) =< 1.2 X ULN
* Total bilirubin =< 1.5 X ULN (may not have abnormalities in both bilirubin and transaminases)
* Alanine amino transferase (ALT) and aspartate aminotransferase (AST) =< 2.5 X ULN (may not have abnormalities in both bilirubin and transaminases)
* Serum creatinine =< 1.5 mg/dL (133 umol/L)
* Or, if serum creatinine > 1.5 mg/dL: calculated creatinine clearance (ClCR) > 50 mL/min
* Urine Protein to Creatinine Ratio (UPC) < 1
* Able to swallow pills whole and retain oral medication
* A female is eligible to enter and participate in this study if the following apply:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

  * A hysterectomy
  * A bilateral oophorectomy (ovariectomy)
  * A bilateral tubal ligation
  * Is post-menopausal
* Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40pg/mL (< 140 pmol/L)
* Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
* Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment and for 3 months after the completion of treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception; acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:

  * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
  * Oral contraceptive, either combined or progestogen alone
  * Injectable progestogen
  * Implants of levonorgestrel
  * Estrogenic vaginal ring
  * Percutaneous contraceptive patches
  * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
  * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
  * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Female subjects who are lactating must discontinue nursing prior to the first dose of study drug and refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug
* A male is eligible to enter and participate in this study if he and his female sexual partner in the reproductive age group agree to use effective methods of contraception

Exclusion Criteria:

* Prior malignancy:

Subjects with a history of a prior malignancy other than angiosarcoma who have been disease-free for at least 2 years prior to the first dose of study drug and/or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible

* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medications for 3 months prior to first dose of study drug; screening with CNS imaging studies (CT or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases
* Clinically significant gastrointestinal (GI) abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
  * Clinically significant (> 1/2 teaspoon) hemoptysis or gastrointestinal hemorrhage in the past 6 months
* Evidence of active bleeding or bleeding diathesis; recent hemoptysis (>= 1/2 teaspoon of red blood within 8 weeks before first dose of study drug)
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* Left ventricular ejection fraction < 50%
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension (defined as systolic blood pressure [SBP] of >= 140 mmHg or diastolic blood pressure [DBP] of >= 90mmHg); Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry; following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals; at least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement; these three values should be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure; the mean SBP / DBP ratio must be < 140/90 mmHg in order for a subject to be eligible for the study
* Cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months

  * Note: subjects with recent DVT who have been therapeutically coagulated for at least 6 weeks are eligible
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery)
* Evidence of active bleeding or bleeding diathesis; recent hemoptysis (>= ½ teaspoon of red blood within 8 weeks before first dose of study drug)
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels (Note: tumor abutting the vessel is acceptable, but contiguous tumor and vessel is not; CT with contrast is strongly recommended to evaluate such lesions)
* Abnormal serum calcium, magnesium, or potassium levels
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Use of any prohibited medication within the timeframes
* Treatment with any of the following therapies:

  * Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib hydrochloride OR
  * Chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
  * Patients who require chronic use of strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers including but not limited to grapefruit juice
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 (except hemoglobin value) and/or that is progressing in severity, except alopecia
* Previous exposure to pazopanib hydrochloride or a vascular endothelial growth factor receptor (VEGFR) targeted kinase therapy, except for bevacizumab or VEGFR-Trap (Aflibercept)
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-11-03 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, Principal Investigator — Fox Chase Cancer Center
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hollings Cancer Center Medical University of South Carolina, Charleston, South Carolina
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 29
Completed | 22
Not Completed | 7
Not completed — Did not initiate therapy | 3
Not completed — Death | 1
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 66 [30 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: PFS Rate
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. PFS was estimated using the method of Kaplan and Meier.
Time Frame: 3 months
Population: Of the 26 patients who started therapy, response was not evaluable in 8 patients due to lab abnormalities at C1D1 (n=1), consent withdrawal (n=2), toxicity (n=4), and non-compliance (n=1)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
percentage of patients | 54.6 [36.0 to 82.9]

2. Primary Outcome: Response Rate Defined as CR
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Standard estimates of the binomial proportion will be used to estimate and place confidence bounds on the several response rates.
Time Frame: 3 months
Population: 7 of 29 patients were not evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 22
Participants | 0

3. Primary Outcome: Response Rate Defined as Partial Response (PR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Partial Response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Standard estimates of the binomial proportion will be used to estimate and place confidence bounds on the several response rates.
Time Frame: 3 months
Population: 7 of 29 patients were not evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 22
Participants | 1

4. Secondary Outcome: Overall Survival of Patients Treated With Pazopanib Hydrochloride
Description: Estimated using the method of Kaplan and Meier.
Time Frame: Up to 107 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 22
weeks | 69.8 [42.3 to 106.7]

5. Secondary Outcome: Evaluation of Toxicity of Pazopanib Hydrochloride in This Patient Population
Description: Toxicities related/unrelated to study treatment with >10% frequency
Time Frame: Up to 2 years
Population: All patients initially enrolled were followed for toxicities
Measure: Number; unit: toxicities
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 29
toxicities | 189

6. Secondary Outcome: Ability of [F-18] FDG PET/CT as an Imaging Agent in Predicting Efficacy or Early Response as Compared With CT Imaging
Description: Descriptive statistics will include mean, SD, median, minimum, and maximum for continuous variables and the numbers and percentages for categorical variables. Summary statistics for changes in SUVs, tumor to background ratios, lesion size, and comparison scores will be analyzed and presented.
Time Frame: Up to 2 years
Population: No data collected for comparison
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 13/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=29)
anemia (Blood and lymphatic system disorders) | 1 (1)
Bilirubin increase (Investigations) | 2
alanine aminotransferase increase (Investigations) | 4
Aspartate aminotransferase increase (Investigations) | 2
abdominal pain (Gastrointestinal disorders) | 2
low platelet (Blood and lymphatic system disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Death (General disorders) | 1
pericardial effusion (Cardiac disorders) | 2
edema (General disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 1
cardiac arrest/death (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
colitis (Gastrointestinal disorders) | 1
dysphagia (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=29)
Rhinitis (Infections and infestations) | 1
Low hemoglobin (Blood and lymphatic system disorders) | 9
Low absolute neutrophil count (Blood and lymphatic system disorders) | 3
Low white blood cell count (Investigations) | 7
Lymphocyte count decrease (Investigations) | 4
Edema (General disorders) | 3
Hypertension (Vascular disorders) | 14
Ortho-hypotension (Vascular disorders) | 2
Palpitation (Cardiac disorders) | 1
Dizzeness (Nervous system disorders) | 8
Fatigue (General disorders) | 18
Anxiety (Psychiatric disorders) | 1
Chills (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hair color changes (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Pruritis (Skin and subcutaneous tissue disorders) | 1
Palmer-Planter erythrodysesthia syndrome (Immune system disorders) | 1
Hemorrhage (General disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Heart burn (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Anorexia (Gastrointestinal disorders) | 9
Mucositis (Gastrointestinal disorders) | 8
Weight lose (Investigations) | 2
Dysgeusia (Nervous system disorders) | 6
confusion (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 3
Neuropathy-Motor (Nervous system disorders) | 4
Neuropathy-Sensory (Nervous system disorders) | 2
Blurred vision (Nervous system disorders) | 3
Pain (General disorders) | 14
Headache (Nervous system disorders) | 14
Myal-arthralgia (Musculoskeletal and connective tissue disorders) | 6
cough (Respiratory, thoracic and mediastinal disorders) | 7
Nose bleeding (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Hypothyroidism (Endocrine disorders) | 1
Alkaline phosphatase increase (Investigations) | 6
Hyperbilirubinemia (Investigations) | 8
SGOT increase (Investigations) | 10
SGPT increase (Investigations) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Infection without neutropenia (Infections and infestations) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Investigations) | 4
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Elevated creatinine (Investigations) | 4
Urinary tract infection (Renal and urinary disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Transaminitis (Investigations) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT01462630/Prot_SAP_000.pdf